CLINICAL TRIAL: NCT00286702
Title: Does Splinting Prevent Contractures Following Stroke?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Sydney (Other)
Other Study IDs: HEC 01/166
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2006-02-03 (Estimated); Status verified 2006-01

CONDITIONS: Cerebrovascular Accident
Keywords: splints; Occupational Therapy
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Device: hand splint

SUMMARY:
After a stroke, many people develop contracture of the muscles in their affected wrist and hand which leads to a permanently clenched, painful hand. A contracture is often treated by therapists who use hand splinting to prevent it occurring or slow down its progression. Despite their wide use, there has not been research completed to investigate whether or not splinting prevents contracture in people following stroke. In fact, this project will be the first of its kind in the world and is therefore vital to stroke rehabilitation.

The study is a multi-centre, randomised controlled trial that will measure the effect of hand-splinting in two positions on the prevention of contracture, functional use of the hand, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* first ever stroke
* score of <1 on Motor Assessment Scale item 6

Exclusion Criteria:

* comorbidity resulting in previous contracture of the wrist/hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63
Dates: Start 2002-10; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Lannin, BSc(OT), Principal Investigator — University of Western Sydney; Anne Cusick, PhD, Study Chair — University of Western Sydney